CLINICAL TRIAL: NCT02357329
Title: Food Composition and Palatability
Acronym: FCandP
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Prof. Nutrition Sciences, Purdue University
Other Study IDs: 055-0390
Record Dates: First submitted 2014-12-22; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2014-12

CONDITIONS: Fat Taste
Keywords: fat taste; food preference; consumption; free fatty acids
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Taste and hedonic ratings of NEFA: Linoleic acid solutions from 0.005% to 1.58%. Participants swish and spit 10 - 7.5mL solutions.

SUMMARY:
This study will investigate fat taste and if free fatty acids (FFA) in food function as a signal for fat content. FFA are quite unpleasant - the investigators want to measure if the concentration in different foods correlates with hedonic preference. FFA concentration from a variety of foods will be used to determine if people who have greater sensitivity for FFA find foods with higher FFA concentrations less acceptable. Further, this study with determine whether the relationship between fat taste and hedonic food preference is modified by sex and body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Healthy
* Non-smoker

Exclusion Criteria:

* Food allergies
* Inability to detect and identify basic tastes

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: unselected convenience sample
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
NEFA sensitivity (Participants will taste and rate 10 solutions based on intensity) | 1 day
  Participants will taste and rate 10 solutions based on intensity

SECONDARY OUTCOMES:
Food consumption and preference (Participants will answer questions regarding consumption of foods and preference) | 1 day
  Participants will answer questions regarding consumption of foods and preference.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue Univeristy, West Lafayette, Indiana, United States